CLINICAL TRIAL: NCT02023645
Title: The Effects of a Lutein + Zeaxanthin Intervention on Cognitive Function and Neural Efficiency
Brief Title: The Effects of a Carotenoid Intervention on Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Georgia (Other)
Collaborators: Abbott Nutrition (Industry); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Billy R. Hammond, Professor and Principal Investigator, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-10516
Record Dates: First submitted 2013-12-16; First posted 2013-12-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Mild Cognitive Impairment
Keywords: lutein; cognition; neural efficiency; aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active supplement (Experimental): 10 mg lutein + 2 mg zeaxanthin
  Interventions: Dietary Supplement: active supplement
- inert placebo (Placebo Comparator): placebo for comparison
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: active supplement — tablet
  Other Names: FloraGlo lutein
  Arms: Active supplement
Other: placebo — tablet
  Other Names: inert placebo
  Arms: inert placebo

SUMMARY:
Past research suggests that retinal lutein levels are related to cognitive function as measured via behavioral tests. The goal of the present study is to investigate the relationship between lutein and cognitive function in a wider variety of the population (young, healthy adults and older adults), using a wider variety of methods (behavioral testing and neuroimaging).

DETAILED DESCRIPTION:
Past research suggests that retinal lutein levels are related to cognitive function as measured via behavioral tests. The goal of the present study is to investigate the relationship between lutein and cognitive function in a wider variety of the population (young, healthy adults and older adults), using a wider variety of methods (behavioral testing and neuroimaging).

ELIGIBILITY:
Inclusion Criteria:

* visual acuity correctable to 20:40 or better, Snellen notation
* able to swallow a dietary supplement
* free of dementia, characterized by a score of less than 1.5 on the Clinical Dementia Rating Scale

Exclusion Criteria:

* GI conditions that interfere with lipid absorption
* presence of or past diagnosis of age-related macular degeneration
* visual acuity poorer than 20:40, Snellen notation
* has taken lutein, omega-3 fatty acid or fish oil supplements within the last 6 months
* presence of dementia, characterized by a score of 1.5 or greater on the Clinical Dementia Rating Scale

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
macular pigment optical density | 12 months
  optical density of macular pigment layer in central retina, defined in log units of optical density

SECONDARY OUTCOMES:
serum carotenoid levels | 12 months
  serum carotenoids will be measured via high performance liquid chromatography
reaction time | 12-months
  reaction (msec) to a light stimulus
executive function | 12-months
  computerized composite score from computerized battery
short-term memory | 12-months
  composite score from a computerized battery
visual attention | 12-months
  composite score from computerized battery

CONTACTS AND LOCATIONS:
Overall Officials: Billy R Hammond, Ph.D., Principal Investigator — The University of Georgia
Locations (1):
- The University of Georgia, Athens, Georgia, United States

REFERENCES:
- [Derived] Mewborn CM, Lindbergh CA, Hammond BR, Renzi-Hammond LM, Miller LS. The Effects of Lutein and Zeaxanthin Supplementation on Brain Morphology in Older Adults: A Randomized, Controlled Trial. J Aging Res. 2019 Dec 1;2019:3709402. doi: 10.1155/2019/3709402. eCollection 2019. PMID 31871787